CLINICAL TRIAL: NCT01272323
Title: An Optional 1 Year Follow up Study to Evaluate the Continued Efficacy of Cat-PAD in Cat Allergic Subjects Following Challenge to Cat Allergen in an Environmental Exposure Chamber
Brief Title: Cat-PAD Follow on Study
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Cetero Research, San Antonio (Network); Adiga Life Sciences, Inc. (Industry)
Responsible Party: Dr Rod Hafner, VP R&D, Circassia Ltd
Other Study IDs: CP005A
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Cat Allergy; Rhinoconjunctivitis
Keywords: Cat allergy; Rhinoconjunctivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Placebo: Subjects previously randomised to receive placebo in study CP005
  Interventions: Biological: Placebo
- Cat-PAD Group 1: Subjects previously randomised to receive Cat-PAD dose 1 in study CP005
  Interventions: Biological: Cat-PAD Dose 1
- Cat-PAD Group 2: Subjects previously randomised to receive Cat-PAD dose 2 in study CP005
  Interventions: Biological: Cat-PAD Dose 2

INTERVENTIONS:
Biological: Placebo — No further medication to be administered in this study. Intervention refers to treatment received in Study CP005.
  Groups: Placebo
Biological: Cat-PAD Dose 1 — No further medication to be administered in this study. Intervention refers to treatment received in Study CP005.
  Groups: Cat-PAD Group 1
Biological: Cat-PAD Dose 2 — No further medication to be administered in this study. Intervention refers to treatment received in Study CP005.
  Groups: Cat-PAD Group 2

SUMMARY:
Cat allergy is an increasingly prevalent condition, affecting 10-15% of patients with allergic rhinoconjunctivitis and/or asthma.

The purpose of this optional observational follow-on study is to further evaluate rhinoconjunctivitis symptoms on exposure to cat dander in the EEC among subjects who completed all dosing visits in study CP005 approximately one year after the start of treatment.

DETAILED DESCRIPTION:
Subjects who completed all dosing visits and the post treatment challenge (PTC) in study CP005 will be invited to attend the Screening Visit for CP005A. Subjects will attend for 4 visits to the EEC on successive days. Following the last EEC visit a follow-up visit will be performed 3-10 days later.

ELIGIBILITY:
Inclusion Criteria

* Previously randomised in study CP005, completed all treatment visits and the Post Treatment Challenge (PTC).

Exclusion Criteria

* "Partly controlled" and "uncontrolled" asthma
* History of anaphylaxis to cat allergen
* FEV1 of less than 70% of predicted
* Subjects who cannot tolerate baseline challenge in the EEC
* Treatment with beta-blockers,Alpha-adrenoceptor blockers, Tranquillizers or psychoactive drugs
* A history of any significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject previously randomised in study CP005 and completed all dosing visits and the PTC
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Score | 50-54 weeks after the start of treatment in CP005

SECONDARY OUTCOMES:
Total Symptom scores for ocular and nasal symptoms | 50-54 weeks after the start of treatment in CP005

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, MD, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Mississauga, Ontario, Canada